CLINICAL TRIAL: NCT00555737
Title: Performance Evaluation of Capsule Endoscopy in the Diagnosis of Gluten Sensitive Enteropathy
Brief Title: Performance Evaluation of Capsule Endoscopy in the Diagnosis of Gluten Sensitive Enteropathy (MA-23)
Status: Completed | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Corporate Director Clinical Affairs, Given Imaging Ltd.
Other Study IDs: MA-23
Record Dates: First submitted 2007-11-08; First posted 2007-11-09 (Estimated); Last update posted 2019-07-31 (Actual); Status verified 2007-11

CONDITIONS: Celiac Disease
Keywords: Celiac Disease; Capsule Endoscopy; small Bowel Disease
MeSH Terms: conditions — Celiac Disease | interventions — Capsule Endoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Capsule Endoscopy — Given® Diagnostic system with Pillcam SB

SUMMARY:
The purpose of this study is to determine how well capsule endoscopy identifies changes in the small bowel mucosa of celiac disease patients.

DETAILED DESCRIPTION:
Gluten-sensitive enteropathy (GSE), also known as celiac disease, is characterized by abnormal small intestinal mucosa arising as a consequence of an inappropriate inflammatory response to ingested gluten in susceptible individuals.

These changes cause a loss of absorptive capacity which in turn leads to variable degrees of malabsorption. A person suffering from celiac may have symptoms ranging from mild iron deficiency anemia to severe diarrhea and weight loss. Characteristically, removal of gluten from the diet is followed by resolution of the mucosal changes and the symptoms.

Celiac disease is suspected on the basis of clinical signs and symptoms, and is generally confirmed by serological testing and small bowel biopsy. Patients with suspected celiac disease undergo upper GI endoscopy with mucosal biopsy of the duodenum, in order to detect the characteristic histological changes.

Although the main role for endoscopy in GSE is to obtain tissue for histological examination, a variety of endoscopic changes have been described in these patients,such as nodularity of the mucosa and 'scalloping' or loss of the duodenal mucosal folds.

The Given® Diagnostic System can visually investigate the small bowel, producing high-quality images of the mucosa, which might be able to detect villous atrophy and thus could be used in the assessment of patients with GSE. Whereas upper GI endoscopy is invasive, often requires sedation and may be uncomfortable, Capsule Endoscopy is less invasive, convenient to use and does not require sedation.

Capsule Endoscopy could become an important tool for the non-invasive assessment of small bowel mucosa in GSE.

ELIGIBILITY:
Inclusion Criteria:

* Patient age is 18 years or older
* Patient agrees to sign the Informed Consent Form
* Patient has positive celiac serology or negative celiac serology + IgA deficiency and suffers from one or more of the following symptoms and/or abdominal biochemical values:

  1. Chronic diarrhea
  2. Weight loss
  3. Abdominal cramps
  4. History of spontaneous abortion
  5. Iron deficiency anemia
  6. Osteoporosis
  7. Infertility
  8. Hypoalbuminaemia
  9. Low cholesterol
  10. Low prothrombin activity

Exclusion Criteria:

* Patient is known or is suspected to suffer from intestinal obstruction.
* Patient has a cardiac pacemaker or other electro-medical device.
* Patient suffers from severe swallowing disorder or Zenker's diverticulum
* Patient has any condition, which precludes compliance with study and/or device instructions.
* Female patient is pregnant
* Patient suffers from life threatening conditions
* Patient is currently participating in another clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: clinic paitnets with known Gluten sensitivity (Celaic).
Sampling Method: Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2003-11; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
The number of findings identified during the capsule endoscopy or upper GI endoscopy procedure, and which were considered by the investigator as related to the gluten sensitive enteropathy origin | within 14 days of enrollment

SECONDARY OUTCOMES:
Longitudinal extent of villous changes in the small bowel will be evaluated. | within 14 days of enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Roberto de Franchis, MD, Prof., Principal Investigator — Ospedale Maggiore - Policlinico, Milano, Italy
Locations (5):
- University of Massachusetts Memorial Medical Center, Worcester, Massachusetts, United States
- University of Tampere Medical School, Tampere, Finland
- Italy (3):
  - Ospedale Maggiore - Policlinico, Milan
  - Universita Cattolica del Sacro Cuore, Rome
  - San Giovanni A.S. Hospital, Torino